CLINICAL TRIAL: NCT02843659
Title: A Phase II, Randomized, Multi-Center, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of BMS-931699 (Lulizumab) or BMS-986142 in Subjects With Moderate to Severe Primary Sjögren's Syndrome
Brief Title: Proof of Concept Study to Evaluate the Efficacy and Safety of BMS-931699 (Lulizumab) or BMS-986142 in Primary Sjögren's Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to meet protocol objectives
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM128-035; 2016-000101-37 (EudraCT Number)
Record Dates: First submitted 2016-07-08; First posted 2016-07-26 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Sjögren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — lulizumab pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-931699 (Experimental): Subcutaneous weekly injection + daily oral placebo tablets
  Interventions: Drug: BMS-931699; Drug: Placebo
- BMS-986142 (Experimental): Daily oral tablets + subcutaneous placebo (weekly) injection
  Interventions: Drug: BMS-986142; Drug: Placebo
- Placebo (Placebo Comparator): Weekly subcutaneous placebo injection +daily oral placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-931699 — Specified dose on specified days
  Other Names: lulizumab
  Arms: BMS-931699
Drug: BMS-986142 — Specified dose on specified days
  Arms: BMS-986142
Drug: Placebo — Specified dose on specified days

SUMMARY:
The primary objective of this study is to evaluate the efficacy of treatment with either lulizumab or BMS-986142 versus placebo in subjects with moderate to severe primary Sjögren's syndrome as measured by the change from baseline in ESSDAI at Week 12 between active treatment arms (lulizumab or BMS-986142, respectively) and the placebo arm.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects diagnosed or classified as having moderate to severe primary Sjögren's Syndrome based on the 2016 ACR-EULAR Sjögren's Syndrome Classification Criteria for at least 16 weeks prior to screening
* ESSDAI ≥ 5 including disease activity (any score > 0) in at least one of the following domains: Glandular, Articular, Hematological, Biological, Lymphadenopathy
* Positive anti-SS-A/Ro and/or anti-SS-B/La autoantibody
* Unstimulated whole saliva secretion > 0.01 ml/min
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug and must not be pregnant or breastfeeding. Male and female subjects must be willing to adhere to protocol-mandated highly effective contraception for the duration of the study and for the protocol-specified follow up period. Hormone-based contraceptive methods are not permitted

Exclusion Criteria:

* Secondary Sjögren's syndrome or the presence of any other systemic autoimmune disease (eg, RA, SLE, multiple sclerosis, vasculitis)
* Very severe primary Sjögren's syndrome or severe complications of primary Sjögren's syndrome at the time of the screening visit
* Active systemic or latent bacterial (including tuberculosis), viral or fungal infection, evidence of current or chronic Hepatitis B or C infection, or HIV infection
* Any significant concurrent medical condition at the time of screening or baseline visit
* Use of methotrexate, cyclophosphamide, cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil (MMF) or leflunomide within 12 weeks of screening visit
* Previous treatment with biologics therapies either marketed or in development within 6 months prior to screening visit
* Treatment started or an unstable dose of hydroxychloroquine within 8 weeks of screening visit
* Oral corticosteroids > 10 mg/day within 14 days of dosing (Day 1), corticosteroid therapy ≥ 1 mg/kg during the 4 weeks preceding enrollment, or intravenous, intramuscular or intra-articular corticosteroids within 4 weeks of screening visit

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (34):
- United States (17):
  - St Joseph Heritage Healthcare, Fullerton, California
  - Local Institution, Palo Alto, California
  - Local Institution, Sarasota, Florida
  - North Georgia Rheumatology Group, Lawrenceville, Georgia
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Local Institution, Tupelo, Mississippi
  - Arthritis And Osteoporosis Associates, Pa, Freehold, New Jersey
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - Local Institution, Mineola, New York
  - Pmg Research Of Wilmington Llc, Wilmington, North Carolina
  - Paramount Medical Research & Consulting, Llc, Middleburg Heights, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Wexford, Pennsylvania
  - Acme Research, Llc, Orangeburg, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Tekton Research Inc, Austin, Texas
- Local Institution, Camperdown, New South Wales, Australia
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Colombia (3):
  - Local Institution, Bogota, Cundinamarca
  - Local Institution, Bogotá
  - Local Institution, Cali
- Azienda Ospedaliera Universitaria Pisana, Pisa, Italy
- Mexico (4):
  - Local Institution, Mexico City, Distrito Fededral
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mérida, Yucatán
  - Local Institution, Veracruz
- Peru (3):
  - Local Institution, Lima Cercado, Lima region
  - Local Institution, Lima
  - Instituto De Ginecologia Y Reproduccion Inv. Clinical Sac, Lima
- Klinika Reumatologii i Chorob Wewnetrznych, Wroclaw, Poland
- Local Institution, San Juan, Puerto Rico
- Local Institution, Moscow, Russia
- Local Institution, Stellenbosch, Western Cape, South Africa

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 subjects enrolled, 18 subjects were randomized/treated. 15 subjects didn't complete the treatment period. The study was terminated and the remaining 15 randomized subjects who had not yet completed the double-blind period entered the follow-up period. Of the 15 subjects who entered the follow-up period, 12 did not complete the follow-up period
Groups:
- BMS-931699/Lulizumab Injection: (12.5mg/vial, 12.5mg/mL) for subcutaneous (SC)
- BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval): For oral administration, 350 mg
- Placebo: For BMS-986142 50 mg tablet (round) or 150 mg tablet
Period: Overall Study
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Started | 5 | 6 | 7
Completed | 1 | 0 | 2
Not Completed | 4 | 6 | 5
Not completed — Subject Withdrew Consent | 0 | 0 | 1
Not completed — Administrative Reason by Sponsor | 4 | 5 | 4
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (11.34) | 51.2 (8.77) | 52.6 (13.30) | 51.2 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 7 | 18
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 4 | 7 | 15
  Black or African American | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in ESSDAI
Description: The ESSDAI is a clinical index that measures Sjogren's syndrome disease activity. A physician scores the disease activity level of twelve organ-specific domains in 3 or 4 levels according to their severity. For example, for no disease activity the domain score equals 0 and for high disease activity the domain score equals 3 or 4. Each domain is assigned a weight between 1 and 6, and the domain score is multiplied by the domain weight. The sum of the weighted domain scores is the overall score, which can range from 0 to 123. A higher score indicates more disease activity. Change from baseline was computed as the value at Week 24 minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening
Time Frame: At baseline and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Mean Change From Baseline in ESSDAI Scores at Week 4 and Week 8
Description: as for outcome 1
Time Frame: At baseline, week 4 and week 8
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Mean Change From Baseline in ESSPRI Score at Week 4, Week 8, and Week 12.
Description: ESSPRI, also known as EULAR Sjogren's Syndrome Patient Reported Index, measures subjective symptoms of dryness, pain and fatigue. It uses 0-10 numerical scales, one for each domain. The weight of the domains is identical, and the final score is the mean score of the 3 domains.
Time Frame: At baseline, week 4, week 8, and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Proportion of Subjects With a > = 3 Point Improvement From Baseline in ESSDAI at Week 12
Description: as for outcome 1
Time Frame: At week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Proportion of Subjects With Both >= 3 Points Improvement in ESSDAI and >= 1 Point Improvement in ESSPRI From Baseline at Week 12
Description: as for outcome 1
Time Frame: At week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Proportions of Subjects With >=1 Point of Improvement From Baseline in ESSPRI
Description: as for outcome 3
Time Frame: At week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Mean Change in Baseline in ESSPRI Individual Component of Dryness
Description: as for outcome 3
Time Frame: At baseline, week 4, week 8, and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Mean Change in Baseline in ESSPRI Individual Component of Fatigue
Description: as for outcome 3
Time Frame: At baseline, week 4, week 8, and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Mean Change in Baseline in ESSPRI Individual Component of Pain
Description: as for outcome 3
Time Frame: At baseline, week 4, week 8, and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Mean Change From Baseline in Unstimulated Salivary Flow Rate
Description: Serum and saliva biomarkers (collected from samples obtained during unstimulated and stimulated salivary flow assessments) were measured to determine the potential PD effect of BMS-931699 and BMS-986142 on disease-related protein analytes. These assessments included, but were not limited to, the detection of cytokines and other protein analytes by immunoassays and/or mass spectrometry proteomic profiling.
Time Frame: At baseline, week 4, week 8, and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Mean Change From Baseline in Stimulated Salivary Flow Rate
Description: as for outcome 10
Time Frame: At baseline, week 4, week 8, and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Mean Change From Baseline in Ocular Surface Staining
Description: The test was performed by instillation of fluorescein dye and either lissamine green or Rose bengal dye to stain the cornea and conjunctiva, respectively. After instilling the dye, the ocular surface was examined through a slit lamp (biomicroscope).
Time Frame: At baseline, week 4, week 8, and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Mean Change From Baseline in Schrimer's Test
Description: The test (without anaesthesia) was performed by placing a narrow calibrated filter-paper strip in the inferior cul-de-sac of each eye. Aqueous tear production was measured by the length in millimeters that the strip wets during the 5 minute test period
Time Frame: At baseline, week 4, week 8, and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Mean Change From Baseline in the Tear Break-up Time Test
Description: Determined by instilling fluorescein dye and evaluating the stability of the pre-corneal tear film. After several blinks, the tear film is examined using a broad beam of the slit-lamp (biomicroscope) with a cobalt blue filter. The TBUT, defined as the time in seconds between the subjects's last blink and the first appearance of a random dry spot on the corneal surface, is measured 3 times and the mean value is recorded.
Time Frame: At baseline, week 4, week 8, and week 12
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Mean Change From Baseline in Numeric Rating Scale (NRS) for Mouth, Eye and Vaginal Dryness
Description: The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. 0 = No Pain, 1-3 = Mild Pain(nagging, annoying, interfering little with ADLs), 4-6 = Moderate Pain (interferes significantly with ADLs), 7-10 = Severe Pain (disabling; unable to perform ADLs)
Time Frame: At baseline, at week 2, week 4, week 6, week 8, week 10, week 12, and week 18
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Mean Change From Baseline in Subject Global Assessment of Disease Activity (SubGDA)
Description: The subjects overall assessment of disease activity from 0-10 cm VAS scale with 0 being no disease and 10 cm being most severe disease
Time Frame: At baseline, week 2, week 4, week 6, week 8, week 10, week 12, and week 18
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Mean Change Form Baseline in Physician Global Assessment of Disease Activity (phyGDA)
Description: The investigator's or physician's overall assessment of disease activity from 0-10 cm VAS scale with 0 being no disease and 10 cm being most severe disease.
Time Frame: At baseline, week 2, week 4, week 6, week 8, week 10, week 12, and week 18
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Mean Change From Baseline in Short Form-36 (SF-36)
Description: First, precoded numeric values are recoded per the scoring key given in Table 1. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Table 2 lists the items averaged together to create each scale. Items that are left blank(missing data) are not taken into account when calculating the scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered
Time Frame: At baseline, week 4, week 8, week 12, and week 18
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Mean Change From Baseline in Female Sexual Function Index (FSFI)
Description: The Female Sexual Function Index (FSFI), a 19-item questionnaire, has been developed as a brief, multidimensional self-report instrument for assessing the key dimensions of sexual function in women
Time Frame: At baseline, week 4, week 8, week 12, and week 18
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Mean Change From Baseline in Work Participation and Activity Impairment Questionnaire (WPAI)
Description: Affords calculation of 4 scales to measure the impact of IBD on different domains of impairment in work or other activities: absenteeism, presenteeism (impairment at work), productivity loss (overall work impairment), activity impairment
Time Frame: At baseline, week 4, week 8, week 12, and week 18
Population: The study was terminated and data is not reported for privacy reasons
Arm/Group | BMS-931699/Lulizumab Injection | BMS-986142 50 mg Tablet (Round) or 150 mg Tablet (Oval) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Groups:
- Placebo: Subjects received subcutaneous (SC) injection of placebo matched to 12.5 milligram (mg) lulizumab (BMS-931699) weekly (QW) and oral tablets of placebo matched to 350 mg BMS-986142 once daily (QD) for 12 weeks.
- Lulizumab (BMS-931699) 12.5mg QW: Subjects received SC injection of 12.5 mg lulizumab (BMS-931699) QW and oral tablets of placebo matched to 350 mg BMS-986142 QD for 12 weeks.
- BMS-986142 350 mg QD: Subjects received oral tablets of 350 mg BMS-986142 QD and placebo matched to SC injection of 12.5 mg lulizumab (BMS-931699) QW for 12 weeks.
Arm/Group | Placebo | Lulizumab (BMS-931699) 12.5mg QW | BMS-986142 350 mg QD
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 1/6
Other Adverse Events (participants affected / at risk) | 2/7 | 4/5 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | Lulizumab (BMS-931699) 12.5mg QW (N=5) | BMS-986142 350 mg QD (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | Lulizumab (BMS-931699) 12.5mg QW (N=5) | BMS-986142 350 mg QD (N=6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Anticoagulation drug level above therapeutic (General disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT02843659/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT02843659/SAP_001.pdf